CLINICAL TRIAL: NCT05370625
Title: A Multicentric, Randomized, Placebo-controlled, Double-blind Study to Assess the Effect of TOTUM-854 on Blood Pressure in Subjects With Moderately Elevated Blood Pressure
Brief Title: To Assess TOTUM-854 on Blood Pressure in Subjects With Moderately Elevated Blood Pressure
Acronym: INSIGHT-2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Valbiotis (Industry)
Collaborators: BioTeSys GmbH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: VCT-012; BTS1815/21 (Other: Biotesys)
Record Dates: First submitted 2022-05-06; First posted 2022-05-11 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-07

CONDITIONS: Elevated Blood Pressure
Keywords: Dietary supplement; Plant extracts
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Totum-854 (Experimental): 2.65-g dose of Totum-854 dietary supplement, a mix of 6 plant extracts. Five capsules per day to consume orally in two intakes Other names: active product
  Interventions: Dietary Supplement: Totum-854
- Placebo (Placebo Comparator): Five capsules per day to consume orally in two intakes
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Totum-854 — To compare Totum-854 with Placebo on blood pressure
  Other Names: Active product
  Arms: Totum-854
Dietary Supplement: Placebo — Five capsules per day to consume orally in two intakes
  Other Names: Comparator product
  Arms: Placebo

SUMMARY:
The main objective of the study will be to compare the efficacy of a 2.65 g/day dose of TOTUM-854 versus placebo in decreasing SBP in subjects with high-normal blood pressure and Grade I hypertension following 12 weeks of daily intake.

ELIGIBILITY:
Main Inclusion Criteria:

* Office Systolic Blood Pressure between 130 and 159 mmHg and Diastolic Blood Pressure < 100 mmHg
* Body Mass Index (BMI) between 18.5 and 35 kg/m²
* Weight stable within ± 5 % in the last three months
* No significant change in food habits or in physical activity in the 3 months prior to randomization and agreeing to keep them unchanged throughout the study

Main Exclusion Criteria:

* Known or suspected secondary hypertension
* Known hypertensive retinopathy and/or hypertensive encephalopathy;
* History of spontaneous or drug-induced angioedema;
* Clinically significant valvular heart disease or severe aortic stenosis
* History of acute coronary syndrome (non-ST elevation myocardial infarction, ST elevation myocardial infarction, and unstable angina pectoris), stroke, or transient ischemic attack within 6 months prior to screening
* Suffering from a severe chronic disease or gastrointestinal disorders found to be inconsistent with the conduct of the study by the investigator

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2022-05-30 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Systolic Blood Pressure at V4 | V4 (12 weeks of intervention)
  Automated Office Blood Pressure (in mmHg), TOTUM-854 vs placebo

SECONDARY OUTCOMES:
Evolution of Systolic Blood Pressure | V0 (inclusion), V2 (4 weeks of intervention), V3 (8 weeks), V4 (12 weeks)
  Automated Office Blood Pressure (in mmHg), TOTUM-854 vs placebo
Evolution of Diastolic Blood Pressure | V0 (inclusion), V2 (4 weeks of intervention), V3 (8 weeks), V4 (12 weeks)
  Automated Office Blood Pressure (in mmHg), TOTUM-854 vs placebo
Evolution of fasting blood glycemia | V0 (inclusion), V2 (4 weeks of intervention), V3 (8 weeks), V4 (12 weeks)
  Glycemia (in mg/dL), TOTUM-854 vs placebo
Evolution of the fasting blood concentration of triglycerides | V0 (inclusion), V2 (4 weeks of intervention), V3 (8 weeks), V4 (12 weeks)
  Triglycerides (in g/L), TOTUM-854 vs placebo
Evolution of the fasting blood concentration of total cholesterol | V0 (inclusion), V2 (4 weeks of intervention), V3 (8 weeks), V4 (12 weeks)
  Total cholesterol (in g/L), TOTUM-854 vs placebo
Evolution of the fasting blood concentration of HDL cholesterol | V0 (inclusion), V2 (4 weeks of intervention), V3 (8 weeks), V4 (12 weeks)
  HDL cholesterol (in g/L), TOTUM-854 vs placebo
Evolution of the fasting blood concentration of non-HDL cholesterol | V0 (inclusion), V2 (4 weeks of intervention), V3 (8 weeks), V4 (12 weeks)
  non-HDL cholesterol (in g/L), TOTUM-854 vs placebo
Evolution of the fasting blood concentration of LDL cholesterol | V0 (inclusion), V2 (4 weeks of intervention), V3 (8 weeks), V4 (12 weeks)
  LDL cholesterol (in g/L, Friedewald method), TOTUM-854 vs placebo
Evolution of fasting blood concentration of hsCRP | V0 (inclusion), V2 (4 weeks of intervention), V3 (8 weeks), V4 (12 weeks)
  hsCRP (in mg/L), TOTUM-854 vs placebo
Evolution of body weight | V0 (inclusion), V2 (4 weeks of intervention), V3 (8 weeks), V4 (12 weeks)
  Body weight (in kg), TOTUM-854 vs placebo
Evolution of waist circumference | V0 (inclusion), V2 (4 weeks of intervention), V3 (8 weeks), V4 (12 weeks)
  Waist circumference (in cm), TOTUM-854 vs placebo
Evolution of hip circumference | V0 (inclusion), V2 (4 weeks of intervention), V3 (8 weeks), V4 (12 weeks)
  Hip circumference (in cm), TOTUM-854 vs placebo
Evolution of waist hip Ratio | V0 (inclusion), V2 (4 weeks of intervention), V3 (8 weeks), V4 (12 weeks)
  Waist Hip Ratio, TOTUM-854 vs placebo
Evolution of cardiovascular disease risk | V0 (inclusion), V2 (4 weeks of intervention), V3 (8 weeks), V4 (12 weeks)
  Systematic Coronary Risk Estimation value from heartscore calculator, TOTUM-854 vs placebo
Delay of occurence of pharmacological treatment requirement for hypertension from V1 | V1 (randomisation), V2 (4 weeks of intervention), V3 (8 weeks), V4 (12 weeks)
  Dealy between V1 and the date at which the investigator will decide to withdraw the subject from the study because he needs a pharmacological treatment to treat his hypertension, TOTUM-854 vs placebo

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Menzel, MD, Principal Investigator — BioTeSys GmbH
Locations (1):
- BioTeSys, Esslingen am Neckar, Germany